CLINICAL TRIAL: NCT06206746
Title: A Prospective, Multicenter, Randomized, Pivotal Study of the May Health System in Transvaginal Ablation of Ovarian Tissue Under Ultrasound Guidance in Women With Infertility Due to Polycystic Ovary Syndrome
Brief Title: The REBALANCE Study - a Prospective, Multicenter, Randomized, Pivotal Study of the May Health System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: May Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR003
Record Dates: First submitted 2023-12-12; First posted 2024-01-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Polycystic Ovary Syndrome; Infertility, Female
Keywords: PCOS; Infertility related to PCOS; Ovulation restoration
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility, Female

STUDY DESIGN:
Intervention Model Description: Control arm has the option to crossover to receive the May Health procedure after completion of the 3 month primary endpoint visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Device arm (Experimental): May Health procedure performed with the use of the May Health system intended for transvaginal ablation of ovarian tissue under ultrasound visualization in women with infertility due to Polycystic Ovary Syndrome.
  Interventions: Device: May Health System
- Control arm (No Intervention): No fertility medication. Crossover participants who choose to crossover after the 3 month follow up visit will restart follow up as per the Device arm.

INTERVENTIONS:
Device: May Health System — The intervention includes the short-term use of the May Health System, which is comprised of three elements: (1) the May Health Needle-Catheter Ablation Device (NCAD) (the Device) a 16 gauge echogenic needle including a bipolar temperature-controlled RF ablation catheter which is clipped and secured onto a vaginal ultrasound probe; (2) the May Health Adapter which is clipped onto the ultrasound probe; and (3) the May Health Generator: a bipolar radiofrequency (RF) ablation platform utilizing the single use May Health NCAD for ovarian tissue ablation. Once the patient is under conscious sedation, the physician guides the May Health system transvaginally with the use of a transvaginal ultrasound. Once the May Health device is safely and securely positioned, the physician will deliver radio frequency energy inside the ovary in order to ablate the tissue.
  Arms: Device arm

SUMMARY:
A Prospective, Multicenter, Randomized, Pivotal Study of the May Health System in Transvaginal Ablation of Ovarian Tissue under Ultrasound Guidance in Women with Infertility due to Polycystic Ovary Syndrome

DETAILED DESCRIPTION:
The objective of the study is to provide evidence for the safety and effectiveness of the May Health System in transvaginal ablation of ovarian tissue under transvaginal ultrasound guidance to restore ovulation in women with infertility due to polycystic ovary syndrome (PCOS) who have not responded to first-line ovulation induction treatment or are contraindicated for or decline such treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 to ≤ 40 years
2. Infertility associated with oligo- or anovulation, AND EITHER:

   2.1 Ultrasonographic evidence of PCOS (ovarian volume ≥ 10 mL and/or ovarian antral follicle count per ovary ≥ 20) OR

   2.2 Evidence of hyperandrogenemia: either clinical (hirsutism defined as modified Ferriman-Gallwey (mFG) level ≥ 4-6 depending on ethnicity) or biochemical (raised serum concentration of androgens, testosterone ≥ 2.5 nmol/L, or FAI > 4)
3. At least one ovary with ovarian volume ≥ 10.0 mL and < 28.0 mL
4. Ovarian accessibility: determined by ability to bring transvaginal ultrasound transducer into close proximity to at least one ovary. (Note: In the situation where only one ovary is appropriately sized according to the preceding criterion, then this requirement applies to the qualifying ovary.)
5. At least one patent fallopian tube and normal uterine cavity as determined by sonohysterogram, hysterosalpingogram, or hysteroscopy/laparoscopy within the last 3 years
6. Has not responded to first-line ovulation induction treatment or is contraindicated for, or declines, such treatment
7. Currently seeking immediate fertility
8. Willing to comply with Clinical Investigation Plan-specified follow-up evaluations
9. Ability to understand study requirements and has sufficient fluency in one of the approved written translations of the Patient Information and Informed consent form
10. Signed informed consent

Exclusion Criteria:

1. Currently pregnant
2. BMI > 40
3. Marked hyperandrogenism (total serum testosterone ≥ 4.5 nmol/L or 130ng/dL)
4. Poor glycemic level control defined as glycohemoglobin (HbA1c) level > 6.5%
5. Bleeding disorders, such as von Willebrand disease, thrombocytopenia, current use of anticoagulation medication, etc.
6. Active genital or urinary tract infection at the time of the procedure
7. Patient with known or suspected periovarian adhesions
8. Previous ovarian surgery (e.g. ovarian drilling, ovarian cysts surgery, or endometriosis surgery on the ovary)
9. Transvaginal ultrasound transducer cannot be brought into proximity of at least one ovary
10. Presence of a pathologic cyst (i.e. endometrioma, dermoid, etc.) of any size, or a follicle, or functional cyst >15 mm on transvaginal ultrasound in ovary to be treated
11. Received > 2 cycles of treatment with gonadotropins for ovarian stimulation without a resulting pregnancy (excludes human chorionic gonadotropin (hCG) trigger injection)
12. Contraindicated to or known previous reaction to anesthesia or sedation regimen
13. Patient not willing to stop all concomitant first-line ovulation induction treatment (clomiphene citrate, letrozole, as well as metformin unless metformin is required for glycemic control) until the 3-month endpoint is reached
14. Male partner's total motile sperm count (TMSC) < 10 million or not available (unless participant is planning donor sperm IUI)
15. Patient is currently participating in another investigational drug or device study that clinically interferes with the endpoints of this study
16. Known or suspected gynecological malignancy
17. General health condition or systemic disease that may contribute to anovulation, infertility, or represent in the opinion of the investigator, a potential increased risk associated with the May Health system

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 195 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Ovulation occurrence | 3 month follow-up
  Occurrence of at least one (1) ovulation
Adverse event collection | Day 0 through 36 month visit
  Adverse events will be collected between and at each study visit after randomization and throughout the duration of the study and analyzed for seriousness, severity, relatedness to the device and/or the procedure, and whether anticipated

SECONDARY OUTCOMES:
Cumulative ovulation rate at 6 months without 1st-line medication | Device arm and Crossover at 6 month visit
  Cumulative ovulation rate at 6 months, without 1st line medication restarted ≥ 3 months post-procedure
Cumulative ovulation rate at 6 months with 1st-line | Device arm and Crossover at 6 month visit
  Cumulative ovulation rate at 6 months, with 1st line medication restarted ≥ 3 months post-procedure
Time to ovulation | Baseline for the control group is day of randomization to the date of first ovulation. Baseline for the treatment group is day of procedure to the date of first ovulation
  Between baseline and 3-month follow-up with weekly assessment
Documented pregnancy | Control Arm, Device Arm, and Crossover group: from baseline to 30 Day, 3 Month; Device Arm and Crossover group only: 6 Month, 12 Month, 24 Month, 36 Month
  Documented pregnancy at any point during the study (participant reported or medical record)
Hormone serum concentrations | Baseline through 36 month visit
  Anti-Müllerian hormone (AMH) serum concentration (ng/mL); Androstenedione serum concentration (ng/dL); Sex Hormone Binding Globulin (SHBG) (nmol/L); Free Androgen Index (FAI)
Pain level after procedure | Device arm and Crossover - Baseline through 7 day visit
  Measured by Visual Analog Scale (VAS) [ranked from 0 (no pain) to 10 (worst pain)], immediately after procedure completion, prior to discharge, 1-, and 7-day follow-up as well as baseline pain level reported by the participant during menstruation as reference
Performance of activities of daily living | Device arm and Crossover: baseline, 24 hours post procedure, D7
  Received score from activities of daily living (ADL)
Procedure times | Device arm and Crossover at Day 0
  Includes pre-treatment, treatment, and post-treatment
Time to discharge | Device arm and Crossover at Day 0
  Defined as time from end-of-procedure until participant meets all conditions to be discharged from Post Anesthesia Care Unit (PACU)
Modified Post Anaesthetic Discharge Scoring System (PADSS) | Device arm and Crossover at 1 hour, 2 hour post procedure
  The Modified Post Anesthetic Discharge Scoring System (PADSS) score is completed after the procedure. The score evaluates whether the participant is safe to go home after anesthesia. It scores 0-2 points in each category (vital signs, activity, nausea/vomiting, pain, bleeding, intake/output), for a maximum score of 10. Discharge can occur with a score of 9 or more and a vital signs score of 2.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Hansen, MD, PhD, Principal Investigator — Oklahoma University Health Sciences Center; Anuja Dokras, MD, PhD, Principal Investigator — Penn Fertility Care
Locations (22):
- United States (22):
  - Bloom Reproductive Institute, PLLC, Scottsdale, Arizona
  - HRC Fertility - Encino, Encino, California
  - UCSF Center for Reproductive Health, San Francisco, California
  - University of South Florida, Tampa, Florida
  - The IVF Center, Winter Park, Florida
  - SIU School of Medicine, Reproductive Endocrinology & Infertility Center, Springfield, Illinois
  - University of Iowa Health Care, Iowa City, Iowa
  - Cypress Medical Research Center, Wichita, Kansas
  - Johns Hopkins Fertility Center, Lutherville, Maryland
  - IVF Michigan, P.C., Bloomfield Hills, Michigan
  - Washington University Fertility and Reproductive Medicine Center, St Louis, Missouri
  - University Reproductive Associates, PC, Hasbrouck Heights, New Jersey
  - University of Rochester, Strong Fertility Center, Rochester, New York
  - Reach Fertility, Charlotte, North Carolina
  - UNC Fertility, Raleigh, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State College of Medicine, Hershey, Pennsylvania
  - Penn Fertility Care, Philadelphia, Pennsylvania
  - Prisma Health - Upstate, Greenville, South Carolina
  - UT Health San Antonio, San Antonio, Texas
  - Baylor Scott & White Medical Center, Temple, Texas
  - UW Health Generations Fertility Care, Middleton, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after deidentification (text, tables, figures and appendices) in annual clinical study report
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Annually, beginning 3 months following FDA submission of annual report, ending 6 months after final report.
Access Criteria: Investigators participating in the study who have been approved by an institutional review board.